CLINICAL TRIAL: NCT02138136
Title: A Multicentre, Long-term Safety, Efficacy, and Pharmacokinetics Study of Lubiprostone in Paediatric Subjects Aged ≥ 6 Years to < 18 Years With Functional Constipation
Brief Title: Lubiprostone for Children With Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sucampo Pharma Americas, LLC (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAG-0211PFC-11S1; 2013-004384-31 (EudraCT Number)
Record Dates: First submitted 2014-05-06; First posted 2014-05-14 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Constipation - Functional
MeSH Terms: interventions — Lubiprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lubiprostone (Experimental): Participants receive lubiprostone twice daily
  Participants must have completed the entire 12-week treatment period during the preceding study. Those who received 12 mcg twice daily (BID) continued to receive 12 mcg, those who received 24 mcg BID continued with that dose.Those of the placebo arm in the previous study weighing less than 50 kg received 12 mcg BID and over 50 kg received 24 mcg BID during this study.
  Interventions: Drug: Lubiprostone

INTERVENTIONS:
Drug: Lubiprostone — 12 or 24 mcg soft capsules for oral administration
  Other Names: Amitiza®

SUMMARY:
This study is for children with constipation.

Children who completed 3 months of treatment in the earlier study (NCT02042183):

* were invited to participate
* will receive lubiprostone for 9 more months
* will see if lubiprostone safely relieves their constipation if taken for a whole year

ELIGIBILITY:
Inclusion Criteria:

* Has completed the 3-month placebo-controlled study (NCT02042183)
* Will continue to abstain from taking concomitant medication (prescribed or over-the-counter) that affects gastrointestinal motility

Exclusion Criteria:

* Has untreated faecal impaction at the time of rolling over into study
* Has significant change in medical status, newly diagnosed and uncontrolled cardiovascular, liver or lung disease, neurologic or psychiatric disorder, or other systemic disease
* Has demonstrated non-compliance with study protocol during the 3-month placebo-controlled study (NCT02042183)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 419 (Actual)
Dates: Start 2014-02-26 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (85):
- United States (67):
  - University of South Alabama Women's and Children's Hospital, Mobile, Alabama
  - Arizona Children's Center at Maricopa Medical Center, Phoenix, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Northwest Arkansas Pediatric Clinic, Fayetteville, Arkansas
  - Arkansas Childrens Hospital Research Institute, Little Rock, Arkansas
  - WCCT Global, Costa Mesa, California
  - Loma Linda University Health Care, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - MCB Clinical Research, Colorado Springs, Colorado
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Emmerson Clinical Research, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Palmetto Professional Research, Hialeah, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - Savin Medical Group Research Center, Miami Lakes, Florida
  - Nemours Childrens Clinic, Pensacola, Florida
  - Children's Center for Digestive Health Care/GI Care for Kids, Atlanta, Georgia
  - Methodist Medical Center, Peoria, Illinois
  - PediaResearch, LLC - Newburgh, Newburgh, Indiana
  - UnityPoint Health Des Moines/ Blank Children's Clinic, Des Moines, Iowa
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Heartland Research Associates, Wichita, Kansas
  - University of Louisville Research Foundation Inc. Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - PediaResearch, LLC - Owensboro, Owensboro, Kentucky
  - Willis-Knighton Physician Network, Shreveport, Louisiana
  - Virgo-Carter Pediatrics, Silver Spring, Maryland
  - Gastrointestinal Associates, PA, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Pioneer Clinical Research, Bellevue, Nebraska
  - Smart Medical Research, Inc., Jackson Heights, New York
  - NY Presbyterian Weill Cornell, New York, New York
  - Morgan Stanley Children's Hospital of New York Presbyterian, New York, New York
  - PriMed Clinical Research, Beavercreek, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cyn3rgy Research, Gresham, Oregon
  - Square-1 Clinical Research, Inc., Erie, Pennsylvania
  - St. Christopher's Hospital for Children Drexel University, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh UPMC, Pittsburgh, Pennsylvania
  - AAPRI Clinical Research, Warwick, Rhode Island
  - Coastal Pediatric Associates - James Island, Charleston, South Carolina
  - Coastal Clinical Research, Charleston, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Coastal Pediatrics Associates - Mount Pleasant, Mt. Pleasant, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - The Jackson Clinic, P.C., Jackson, Tennessee
  - 3rd Coast Research Associates, Corpus Christi, Texas
  - Childrens Medical Center Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Envision Clinical Research, LLC, Laredo, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Bridgerland Clinical Research, Logan, Utah
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Wee Care Pediatrics, Syracuse, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia
  - INOVA Pediatric Digestive Diseases Center, Fairfax, Virginia
  - Pediatric Gastroenterology Carilion Medical Center, Roanoke, Virginia
  - Northwest Clinicial Research Center, Bellevue, Washington
  - Zain Research LLC, Richland, Washington
  - MultiCare Health System Institute for Research and Innovation, Tacoma, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (2):
  - Universitair Kinderziekenhuis Brussel, Brussels
  - CHC - Clinique Saint-Joseph, Montegnée
- Sainte Justine University Health Center, Montreal, Canada
- CHU-Bordeaux, Bordeaux, France
- Netherlands (4):
  - Emma Children's Hospital, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Maasstad Hospital Rotterdam, Rotterdam
  - Isala Klinieken, Zwolle
- Poland (6):
  - Medical University of Bialystok, Bialystok
  - Szpital Uniwersytecki, Bydgoszcz
  - Szpital Pediatryczny ICZMP, Lodz
  - Gabinet Lekarski Bartosc Korczowski, Rzeszów
  - Przychodnia Specjalistyczna PROSEN, Warsaw
  - Children's Memorial Health Institute, Warsaw
- United Kingdom (4):
  - Darlington Memorial Hospital, Darlington
  - Royal London Hospital, London
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - Sheffield Children Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benninga MA, Hussain SZ, Sood MR, Nurko S, Hyman P, Clifford RA, O'Gorman M, Losch-Beridon T, Mareya S, Lichtlen P, Di Lorenzo C. Lubiprostone for Pediatric Functional Constipation: Randomized, Controlled, Double-Blind Study With Long-term Extension. Clin Gastroenterol Hepatol. 2022 Mar;20(3):602-610.e5. doi: 10.1016/j.cgh.2021.04.005. Epub 2021 Apr 7. PMID 33838349

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed the 3-month placebo-controlled study (NCT02042183) were invited to enroll in this safety extension study lasting an additional 9 months.
Groups:
- All Participants: Participants received lubiprostone
Period: Overall Study
Arm/Group | All Participants
Started | 419
Safety Analysis Set | 419
Modified Intent to Treat (mITT) (One participant excluded for serious compliance issues with potential data integrity impact) | 418
Completed | 280
Not Completed | 139
Not completed — Protocol Violation | 4
Not completed — Physician Decision | 7
Not completed — Lack of Efficacy | 35
Not completed — Pregnancy | 2
Not completed — Adverse Event | 18
Not completed — Withdrawal by Subject | 36
Not completed — Lost to Follow-up | 32
Not completed — Withdrawn by Sponsor | 5

BASELINE CHARACTERISTICS:
Population: mITT population
Groups:
- All Participants: Participants receive lubiprostone
Arm/Group | All Participants
Number analyzed (Participants) | 418
Age, Customized [Count of Participants; unit: Participants]
  6-17 years of age | 418
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229
  Male | 189
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 36
  Belgium | 2
  United States | 359
  Poland | 10
  United Kingdom | 10
  France | 1

OUTCOME MEASURES:

1. Primary Outcome: Median Number of Observed Weekly Spontaneous Bowel Movements (SBM) Per Month
Description: Spontaneous bowel movements are defined as bowel movements without the aid of drugs.
Time Frame: within 9 months
Population: mITT with evaluable data at the given time point
Measure: Median (Full Range); unit: Weekly SBMs
Arm/Group | All Participants
Number analyzed (Participants) | 418
Weekly SBMs
  Month 1: number analyzed (Participants) | 415
  Month 1 | 2.66 [0.00 to 15.00]
  Month 2: number analyzed (Participants) | 391
  Month 2 | 2.75 [0.00 to 14.73]
  Month 3: number analyzed (Participants) | 373
  Month 3 | 2.70 [0.00 to 18.38]
  Month 4: number analyzed (Participants) | 344
  Month 4 | 2.75 [0.00 to 12.83]
  Month 5: number analyzed (Participants) | 327
  Month 5 | 2.74 [0.00 to 14.00]
  Month 6: number analyzed (Participants) | 313
  Month 6 | 2.50 [0.00 to 7.75]
  Month 7: number analyzed (Participants) | 303
  Month 7 | 2.63 [0.00 to 12.11]
  Month 8: number analyzed (Participants) | 291
  Month 8 | 2.63 [0.00 to 11.00]
  Month 9: number analyzed (Participants) | 269
  Month 9 | 2.50 [0.00 to 10.75]

2. Other Pre Specified Outcome: Median Monthly Score on a 5-point Straining Scale Associated With Observed SBMs
Description: Straining during observed SBMs is rated on a 5-point scale where 1=no straining and 5=extreme straining. A higher value is worse.
Time Frame: within 9 months
Population: mITT with evaluable data at the given time point
Measure: Median (Full Range); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 418
score on a scale
  Month 1: number analyzed (Participants) | 404
  Month 1 | 1.19 [0.00 to 4.00]
  Month 2: number analyzed (Participants) | 373
  Month 2 | 1.25 [0.00 to 4.00]
  Month 3: number analyzed (Participants) | 361
  Month 3 | 1.14 [0.00 to 4.00]
  Month 4: number analyzed (Participants) | 334
  Month 4 | 1.17 [0.00 to 4.00]
  Month 5: number analyzed (Participants) | 314
  Month 5 | 1.19 [0.00 to 4.00]
  Month 6: number analyzed (Participants) | 299
  Month 6 | 1.13 [0.00 to 3.90]
  Month 7: number analyzed (Participants) | 286
  Month 7 | 1.00 [0.00 to 4.00]
  Month 8: number analyzed (Participants) | 271
  Month 8 | 1.00 [0.00 to 4.00]
  Month 9: number analyzed (Participants) | 256
  Month 9 | 1.00 [0.00 to 4.00]

3. Other Pre Specified Outcome: Median Monthly Score on a Stool Consistency Scale Associated With Observed SBMs
Description: Stool consistency is rated on a 5-Point Stool Consistency Scale, where 1=normal and 5=very hard. Higher scores mean a worse outcome.
Time Frame: within 9 months
Population: mITT with evaluable data at the given time point
Measure: Median (Full Range); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 418
score on a scale
  Month 1: number analyzed (Participants) | 404
  Month 1 | 2.80 [1.00 to 5.00]
  Month 2: number analyzed (Participants) | 374
  Month 2 | 2.75 [1.00 to 5.00]
  Month 3: number analyzed (Participants) | 361
  Month 3 | 2.78 [1.00 to 5.00]
  Month 4: number analyzed (Participants) | 334
  Month 4 | 2.78 [1.00 to 5.00]
  Month 5: number analyzed (Participants) | 314
  Month 5 | 2.83 [1.00 to 4.50]
  Month 6: number analyzed (Participants) | 299
  Month 6 | 2.83 [1.17 to 4.50]
  Month 7: number analyzed (Participants) | 286
  Month 7 | 2.87 [1.00 to 5.00]
  Month 8: number analyzed (Participants) | 271
  Month 8 | 2.90 [1.00 to 4.64]
  Month 9: number analyzed (Participants) | 256
  Month 9 | 2.89 [1.00 to 5.00]

4. Other Pre Specified Outcome: Median Monthly Score on a 4-point Pain Scale for Observed Abdominal Pain
Description: Abdominal pain was rated on a scale from 1 (no pain) to 4 (very severe pain). A higher score means a worse outcome.
Time Frame: within 9 months
Population: mITT with evaluable data at the given time point
Measure: Median (Full Range); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 418
score on a scale
  Month 1: number analyzed (Participants) | 416
  Month 1 | 1.00 [0.00 to 4.00]
  Month 2: number analyzed (Participants) | 391
  Month 2 | 0.99 [0.00 to 4.00]
  Month 3: number analyzed (Participants) | 371
  Month 3 | 0.90 [0.00 to 4.00]
  Month 4: number analyzed (Participants) | 352
  Month 4 | 0.85 [0.00 to 4.00]
  Month 5: number analyzed (Participants) | 328
  Month 5 | 0.84 [0.00 to 4.00]
  Month 6: number analyzed (Participants) | 314
  Month 6 | 0.82 [0.00 to 4.00]
  Month 7: number analyzed (Participants) | 306
  Month 7 | 0.75 [0.00 to 4.00]
  Month 8: number analyzed (Participants) | 290
  Month 8 | 0.85 [0.00 to 4.00]
  Month 9: number analyzed (Participants) | 272
  Month 9 | 0.79 [0.00 to 3.81]

ADVERSE EVENTS:
Time Frame: from first open-label dose to last open-label dose plus 7 days (9 months, 7 days)
Description: Only treatment-emergent adverse events (AEs) are reported. Adverse events with onset dates after the administration of the first open-label dose and prior to the last open-label dose plus 7 days are considered treatment-emergent.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/419
Serious Adverse Events (participants affected / at risk) | 13/419
Other Adverse Events (participants affected / at risk) | 147/419
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=419)
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Conversion disorder (Psychiatric disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 2 (2)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=419)
Headache (Nervous system disorders) | 33 (33)
Nausea (Gastrointestinal disorders) | 36 (36)
Vomiting (Gastrointestinal disorders) | 47 (47)
Abdominal pain (Gastrointestinal disorders) | 33 (33)
Diarrhoea (Gastrointestinal disorders) | 27 (27)
Nasopharyngitis (Infections and infestations) | 31 (31)
Upper respiratory tract infection (Infections and infestations) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT02138136/Prot_SAP_000.pdf